CLINICAL TRIAL: NCT06770361
Title: Creation of a Vascular Access Specialist Teams Within an Interventional Vascular Radiology Service: a Retrospective Observational Study
Acronym: ANGIO-ETI
Status: Completed | Type: Observational
Sponsor: Hospital Arnau de Vilanova (Other)
Responsible Party: Principal Investigator, Ferran Padilla Nula, Registred Nurse (RN) and Master of Science (MSc), Hospital Arnau de Vilanova
Other Study IDs: 02/23
Record Dates: First submitted 2024-12-27; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Vascular Access Complication; Nurse; Vascular Access Devices; Nurses
Keywords: Nurse Specialists; Vascular Access Team; Vascular Access Specialist Teams; VAT; VAST

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Hospitalised patients who had undergone an ultrasound-guided catheter cannulation.: Hospitalised patients who had undergone ultrasound-guided catheter cannulation by the vascular access team (VAT) of the Hospital Universitari Arnau de Vilanova (HUAV) of Lleida, integrated in an interventional vascular radiology unit, from 12 September 2017 (day of creation of the unit) until 31 December 2022.

SUMMARY:
A study will be carried out to observe catheters (polyurethane tubes inserted into veins) over a period of five years. The study will look at any problems related to these devices, especially those put in at a specific hospital unit (vascular interventional radiology service) of the Arnau de Vilanova hospital in Lleida (Catalonia, Spain).

DETAILED DESCRIPTION:
Introduction: Vascular Access Specialist Teams (VAST) have been implemented in numerous hospitals worldwide with excellent results. Although these vary in structure and function the purpose is the same in all of them, the improvement in cannulation and comprehensive cures of vascular access devices (VADs) based on the best scientific evidence.

Hypothesis: The creation of a VAST within an Interventional Vascular Radiology (IVR) service reduces the main complications related to VADs and contributes to improving the quality and safety standards necessary in the implantation and treatment of these devices Objective: To describe the creation of a VAST within an IVR service in a second level hospital. In addition, it is expected to analyze the prevalence of VADs placement and success rate, to determine the number of catheter-related bacteremia's and to know the number of failures of VADs cannulated in the EIAV in acute hospitalized patients.

Methodology: Retrospective observational study. A description will be made of the characteristics of the VAST, the implanted VADs and the main associated complications.

Expected results: We expect to describe the structure of a VAST within an IVR service and to analyze the prevalence of VADs placement and success rate, to determine the number of catheter-related bacteremia's and to know the number of failures of VADs cannulated in the VAST in acute hospitalized patients.

Clinical implication: The study will help to improve current VAST and to reduce the difficulties in the creation of future VAST, as well as to clarify the need for these specialized teams, which aim to improve the quality and safety standards necessary for VADs implantation and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Admitted to a hospitalisation unit
* Requiring VAD cannulation for intravenous treatment or due to poor venous access, in accordance with the protocol of insertion criteria of the hospital.

Exclusion Criteria:

- Patients who underwent initial evaluation and cannulation was not attempted are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During the study period, 1,588 consultations were recorded in the unit for VAD cannulation, originating from various hospitalisation units.A non-probabilistic convenience sampling method was employed, and all patients over the age of 18 who were admitted to a hospitalisation unit and required VAD cannulation for intravenous treatment or due to poor venous access were included in the study, in accordance with the hospital's insertion criteria protocol. Patients who underwent the initial assessment but for whom cannulation was not attempted were excluded from the study.Cannulations were performed according to a checklist and with the assistance of ultrasound as a guiding technique.The VAST was created within an IVR service, with specific characteristics and the possibility of being able to channel the VADs in a room with a laminar ventilation system and a fluoroscope arch.
Sampling Method: Non-Probability Sample
Enrollment: 1588 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of complications that result in the malfunction of venous catheters cannulated using the ultrasound-guided technique in an interventional vascular radiology unit, necessitating their removal or replacement. | From date of study entry (day of catheter insertion) to the day of withdrawal from any cause, evaluated up to 111 weeks.
  The present study aims to provide a comprehensive overview of the number of cases in which patients had to undergo catheter removal or replacement due to catheter dysfunction. This dysfunction can be categorised into two distinct types: immediate complications, which include pain, bleeding, haemorrhage, haematoma, difficulty in progressing the guidewire and/or catheter, and arrhythmia, among others; and late complications, which encompass phlebitis, obstruction, extravasation, thrombosis, and infection, to name a few. Furthermore, the list should include the name of complications associated with premature catheter removal, and the rate of complications per 1000 catheter days for catheters cannulated in the unit should be described.

SECONDARY OUTCOMES:
Number of catheter-related bloodstream infections (CRBSI) | From date of study entry (day of catheter insertion) to the day of withdrawal from any cause, evaluated up to 111 weeks.
  The number of catheter-related bloodstream infections (CRBSI) must be described and analysed, as well as the samples and the types of bacteria, viruses or fungi confirmed. The rate of CRBSI per 1000 catheter days in catheters catheterised in the unit must be defined.
Provide the success rate of ultrasound-guided cannulation of vascular access team. | From date of study entry (day of catheter insertion) to the day of withdrawal from any cause, evaluated up to 111 weeks.
  The number of catheters that have had no immediate or late complications and have been able to complete treatment without problems should be provided. In addition, the type of catheter (mini-midline, midline, PICC, etc.) cannulated by the vascular access team and the success rate of each should be described.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Arnau de Vilanova, Lleida, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No